CLINICAL TRIAL: NCT02545322
Title: Image Guided Adaptive Radiotherapy Based on Elastic Image Registration for Improved Tumor Coverage and Reduction of Side Effect in Normal Tissues
Brief Title: Image Guided Adaptive Radiotherapy in the Head-and-neck Region
Acronym: BART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BART 1.1
Record Dates: First submitted 2015-07-29; First posted 2015-09-09 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adaptive Radiotherapy (Experimental): Follow-up CT scans during week 3 and week 5 of Treatment
  Image-guided adaptive Radiotherapy arm:
  Follow-up CT scans are performed on a conventional CT-simulator. Deformable Image Registration between the planning-CT and the follow-up CT (fCT) is done using a dedicated Software package. Delineations for target volumes and organs at risk are transferred to the fCT based on the Deformation vector fields calculated during deformable Image registration. Volumetric changes in target volumes and organs-at-risk are assessed. The initial treatment plan is transferred to the fCT scan. Dosimetric consequences of morphologic changes are analysed with the Focus on target dose coverage for the planning target volume. Adaption and plan re-optimisation are performed.
  Interventions: Radiation: Follow-up CT scans during week 3 and week 5 of treatment

INTERVENTIONS:
Radiation: Follow-up CT scans during week 3 and week 5 of treatment — Scheduled follow-up planning CT scan and re-optimisation of the intensity modulation radiation therapy (IMRT)-based radiotherapy Treatment plan. Dosimetric Evaluation and assessment of morphologic changes.

SUMMARY:
Aim of this study is the clinical evaluation of an image-guided adaptive radiotherapy concept. This involves the adaption of the radiotherapy treatment plan according to changes in tissues and variations in patients position and posture during a radiotherapy treatment course, based on repeat CT scans.

It is investigated, if dosimetric improvements can be achieved using this approach and if the method using the software-package "ReDeform" can be implemented in clinical Routine.

DETAILED DESCRIPTION:
Aim of this study is the clinical evaluation of an image-guided adaptive radiotherapy (ART) concept. This involves the adaption of the radiotherapy treatment plan according to changes in tissues and variations in patients position and posture during a radiotherapy treatment course, based on repeat CT scans.

It is prospectively investigated, if dosimetric improvements can be achieved using this approach and if the method using the software-package "ReDeform" can be implemented in clinical Routine. For that purpose 2 repeat CT scans are acquired during the radiotherapy course (week 3 and week 5 of radiotherapy). The Initial CT scan is "matched" to the follow-up CT-scan by means of deformable image registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histo-pathologically verified malignancies in the head-and-neck without clinical signs of dissemination, who consented in radiotherapy or radio-chemotherapy.

Exclusion Criteria:

* previous radiation therapy for head-and-neck

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin S Kapp, MD, Prof., Principal Investigator — Medical University of Graz

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adaptive Radiotherapy
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adaptive Radiotherapy
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Region of Enrollment [Number; unit: participants]
  Austria | 18

OUTCOME MEASURES:

1. Primary Outcome: Planning Target Volume (PTV) Coverage Parameter D98%
Description: Dose coverage of the planning target volume: Number of participants with a decrease in the planning target volume (PTV) coverage (D98%) above 5%. The Parameter "D98%" denotes the minimum dose to 98% of the volume according to the ICRU (International Commission on Radiation Units & Measurements) Report No. 62. It is a widely accepted classification index for dose coverage.
  The "Planing Target Volume" is a volume, consisting of the clinical target volume and additional safety margins, that should receive a certain radiation dose.
Time Frame: week 5
Measure: Number; unit: participants
Arm/Group | Adaptive Radiotherapy
Number analyzed (Participants) | 15
participants | 7

2. Secondary Outcome: Volumetric Changes
Description: Percent changes in the volume of the Planning Target Volume (PTV). The "Planning Target Volume" is a volume, consisting of the clinical target volume and additional safety margins, that should receive a certain radiation dose. The volumetric changes of the PTV throughout the course of Radiation therapy are evaluated. A significant change in the volume of the PTV (measured in ccm) might be an indicator for possible undesireable dosimetric alterations.
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Adaptive Radiotherapy
Number analyzed (Participants) | 15
percent | -4.3 (5.4)

ADVERSE EVENTS:
Arm/Group | Adaptive Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes